CLINICAL TRIAL: NCT00062179
Title: A Randomized Double Blind Phase II Study of Preoperative Celecoxib/Paclitaxel/Carboplatin for Stage IIIA Non-Small Cell Lung Cancer
Brief Title: Paclitaxel and Carboplatin With or Without Celecoxib Before Surgery in Treating Patients With Stage IIIA Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pharmacia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000304540; UCLA-0208074; NYH-CMC-0902-464; PHARMACIA-COXAON-0509-106
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Celecoxib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paclitaxel/carboplatin/celecoxib (Experimental): Paclitaxel: 225 mg/m2 by 3-hour intravenous infusion Carboplatin: dosed at an AUC of 6 by the Calvert Formula Celecoxib: 400 mg po BID 3 cycles of paclitaxel and carboplatin 21 days apart celecoxib 3-7 days before first dose of chemotherapy
  Interventions: Drug: carboplatin; Drug: celecoxib; Drug: paclitaxel
- paclitaxel/Carboplatin/Placebo (Placebo Comparator): Paclitaxel: 225 mg/m2 by 3-hour intravenous infusion Carboplatin: dosed at an AUC of 6 by the Calvert Formula Placebo 3 cycles of paclitaxel and carboplatin 21 days apart Placebo 3-7 days before first dose of chemotherapy
  Interventions: Drug: carboplatin; Drug: paclitaxel; Other: Placebo

INTERVENTIONS:
Drug: carboplatin — Carboplatin: dosed at an AUC of 6 by the Calvert Formula 3 cycles of carboplatin 21 days apart
Drug: celecoxib — Celecoxib: 400 mg po BID celecoxib 3-7 days before first dose of chemotherapy
  Arms: paclitaxel/carboplatin/celecoxib
Drug: paclitaxel — Paclitaxel: 225 mg/m2 by 3-hour intravenous infusion 3 cycles of paclitaxel 21 days apart
Other: Placebo — placebo 3-7 days before first dose of chemotherapy
  Arms: paclitaxel/Carboplatin/Placebo

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as paclitaxel and carboplatin use different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may increase the effectiveness of a chemotherapy drug by making tumor cells more sensitive to the drug, may stop the growth of tumor cells by stopping blood flow to the tumor, and/or may block the enzymes necessary for tumor cell growth. Giving combination chemotherapy with celecoxib before surgery may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving paclitaxel together with carboplatin followed by surgery works compared to giving paclitaxel together with carboplatin and celecoxib followed by surgery in treating patients with stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the complete pathological response rate and/or minimal residual microscopic disease in patients with stage IIIA non-small cell lung cancer treated with preoperative paclitaxel and carboplatin with vs without celecoxib.
* Compare the clinical response rate in patients treated with these regimens.
* Compare chemotherapy-related toxicity in patients treated with these regimens.
* Compare the time to progression, disease-free survival, and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to use of aspirin for prior cardiovascular disease (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on days 1, 22, and 43. Patients also receive oral celecoxib twice daily beginning on day 1 and continuing until the morning of surgical resection.
* Arm II: Patients receive paclitaxel and carboplatin as in arm I and an oral placebo twice daily beginning on day 1 and continuing until the morning of surgical resection.

In both arms, patients undergo surgical resection and complete mediastinal lymph node dissection within 3-6 weeks after completion of chemotherapy. Patients resume oral celecoxib or placebo twice daily within 28-42 days after surgery and continue until 3 years from the date of randomization in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3-6 months.

PROJECTED ACCRUAL: A total of 110 patients (55 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven non-small cell lung cancer clinical stage IIIA
* Mediastinoscopy positive N2 disease is mandatory
* The disease must be deemed potentially resectable by the thoracic surgeon
* Karnofsky performance status > 80%
* Pulmonary function must be acceptable for surgery according to institutional standards
* Acceptable hepatic, renal and bone marrow function

  * Total serum bilirubin < ULN
  * AST and/or ALT < 2.5x ULN
  * Alkaline phosphatase < 2.5x ULN
  * Serum creatinine < 2.0 mg/mm3
  * White blood cell > 3000/mm3
  * Platelets > 100,000/mm3
* Age 18 or older
* Willingness to abstain from chronic use of NSAIDs (defined as > 7 days of continuous therapy per month OR defined as frequency of > 3 times per week) for the duration of the study. For those patients on NSAIDs prior to study entry, cessation of the drug for 72 hours prior to study entry is required
* Patients on low-dose ASA (<325 mg daily) for prophylaxis of cardiovascular disease prior to study entry may remain on that dose of ASA during this trial
* No anticipated chronic use of steroids. Patients may take the inhaled steroids mometasone or fluticasone if medically indicated

Exclusion Criteria:

* Patients with known hypersensitivity or allergic reactions to COX-2 inhibitors, sulfonamides, NSAIDs, or salicylates
* Hypersensitivity to paclitaxel
* Significant medical or psychiatric illness that would interfere with patient compliance
* Prior malignancy within the last 3 years with the exception of non-melanoma skin cancer
* Receiving other investigational agents during the course of this study or are < 3 weeks from completion of other clinical trial therapy
* Patients with a history of peptic ulcer disease, bleed disorder, irritable bowel disease, inflammatory bowel syndrome, chronic diarrhea or bowel obstruction within 5 years
* Patients receiving enzyme-inducing anticonvulsants are ineligible. Patients who require concomitant therapy with NSAIDs or COX-2 inhibitors
* Patients with any other serious underlying medical condition that would impair the ability of the patient to receive or comply with protocol treatment
* Patients receiving lithium or fluconazole
* Pregnant women or women of childbearing potential that refuse to use effective contraception during the period of chemotherapy.
* Patients with a significant history of unstable cardiovascular disease
* Uncontrolled diabetes mellitus or uncontrolled infection, including HIV or interstitial pneumonia or interstitial fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Rates of complete pathological response and/or minimal residual microscopic disease at 3 years | 3 years

SECONDARY OUTCOMES:
Clinical response at 3 years | 3 years
Difference in time to progression, disease-free survival, and overall survival between Arm I and Arm II at 3 years | 3 years
Toxicity in patients with paclitaxel/carboplatin/celecoxib vs. paclitaxel/carboplatin/placebo

CONTACTS AND LOCATIONS:
Overall Officials: Karen Rickard, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York